CLINICAL TRIAL: NCT01016756
Title: Genetic Analysis of PHACE Syndrome.(PHACE Syndrome is Defined as a Hemangioma Plus One or More of the Following: Brain, Heart, Eye, Sternal or Cerebral Artery Anomalies).
Brief Title: Genetic Analysis of PHACE Syndrome (Hemangioma With Other Congenital Anomalies)
Acronym: PHACE
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Dawn Siegel, Professor, Stanford University
Other Study IDs: PHACE_GENETICS
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: PHACE Syndrome
Keywords: PHACE syndrome; Hemangioma; Coarctation of aorta; Dandy Walker; Brain malformation; Eye anomaly; Sternal malformation; Genetic analysis; Cerebral artery anomaly
MeSH Terms: conditions — Aortic Aneurysm, Giant Congenital; Hemangioma; Aortic Coarctation; Eye Abnormalities

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (4 ml), saliva, buccal swabs and DNA and tissue collection from tissue that would otherwise be discarded after surgery.
Oversight: Data Monitoring Committee: No

SUMMARY:
1. PHACE syndrome(OMIM database number 606519) is the association of a vascular birthmark (hemangioma) on the face along with one or more of the following conditions: congenital heart defects, congenital anomalies of the cerebral arteries,brain, eyes, or sternum.
2. A research study is currently being conducted at the Medical College of Wisconsin (MCW) to investigate if there is an inherited cause of PHACE syndrome.
3. We are hoping that this study will lead to a better understanding of how and why children develop PHACE syndrome.

DETAILED DESCRIPTION:
If you and your child agree to participate in this study, the following will happen:

1. The principal investigator at MCW, or her appointed representative or collaborators at other sites, will review the study protocol and consent form with you and answer any questions- this can be done over the phone.
2. If you choose to participate, the investigator will obtain informed consent for study participation, consent to obtain medical records, and a small amount of logistical information such as address and phone number.
3. Subjects and parents may have a blood draw, saliva sample or buccal swab done.
4. If the subject undergoes surgery for another reason and there is tissue which would otherwise be discarded, we may ask to receive this sample for research purposes.
5. We will request completion of surveys about the individual's medical history as it relates to this condition.
6. The purpose of this study is to promote the understanding of the inheritance of hemangiomas associated with brain, eye and heart anomalies. The DNA obtained from participants are stored in a DNA repository and genetic data bank for current and future research projects related to their genetic disorders. The DNA specimens will be used to map disease-related genes. The principal investigator uses her discretion to decide which investigators will have access to this resource. The analysis of the specimens will vary depending on the investigator and his/her specific protocol.

ELIGIBILITY:
Inclusion Criteria:

* meets the clinical diagnostic criteria for PHACE syndrome.

Exclusion Criteria:

* fails to meet the clinical diagnostic criteria for PHACE syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a facial hemangioma, along with one or more of the following:
  posterior fossa malformation, arterial anomalies, cardiac defects, eye anomalies and sternal anomalies.
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Establish a DNA and tissue bank. | 5 years
Determine candidate genes for PHACE syndrome using a genome-wide approach. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Siegel, MD, Principal Investigator — Stanford University
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Metry D, Heyer G, Hess C, Garzon M, Haggstrom A, Frommelt P, Adams D, Siegel D, Hall K, Powell J, Frieden I, Drolet B; PHACE Syndrome Research Conference. Consensus Statement on Diagnostic Criteria for PHACE Syndrome. Pediatrics. 2009 Nov;124(5):1447-56. doi: 10.1542/peds.2009-0082. Epub 2009 Oct 26. PMID 19858157
- [Background] Metry DW, Haggstrom AN, Drolet BA, Baselga E, Chamlin S, Garzon M, Horii K, Lucky A, Mancini AJ, Newell B, Nopper A, Heyer G, Frieden IJ. A prospective study of PHACE syndrome in infantile hemangiomas: demographic features, clinical findings, and complications. Am J Med Genet A. 2006 May 1;140(9):975-86. doi: 10.1002/ajmg.a.31189. PMID 16575892
- [Background] Frieden IJ, Reese V, Cohen D. PHACE syndrome. The association of posterior fossa brain malformations, hemangiomas, arterial anomalies, coarctation of the aorta and cardiac defects, and eye abnormalities. Arch Dermatol. 1996 Mar;132(3):307-11. doi: 10.1001/archderm.132.3.307. PMID 8607636